CLINICAL TRIAL: NCT02384447
Title: Correlation of the Ultrasound Appearance of the Sciatic Nerve With Its Histologic Appearance in Pathology Specimens Obtained From Patients Undergoing Above Knee Amputation
Brief Title: Comparing the Ultrasound Appearance of the Sciatic Nerve With Its Appearance Under a Microscope
Status: Withdrawn | Type: Observational
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Principal Investigator, Shashi Bhatt, MD, Principal Investigator, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Other Study IDs: UTIRB 0000200125
Record Dates: First submitted 2014-08-07; First posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes
Keywords: above knee amputation; sciatic nerve; ultrasonography; histology
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Amputated extremity for histologic examination of the sciatic nerve.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee Amputation: Patients that are scheduled to undergo above knee amputation due to complications associated with diabetes will be enrolled

SUMMARY:
The investigators are proposing to conduct this study to compare the ultrasonographic appearance of the sciatic nerve with their corresponding histologic architecture. Patients that are scheduled to undergo above knee amputation due to complications associated with diabetes will be enrolled. We intend to do an ultrasound examination of the sciatic nerve at its bifurcation (about 4 inches above the knee). The investigators would mark the area on the skin where the image is obtained. Following surgery we will conduct a histologic examination of the nerve at the same site.

Ultrasound examination is not standard of care, but is a fairly noninvasive procedure and does not add any risk to the subject. Histologic examination of the nerve is also not standard of care, but is conducted on a pathology specimen

ELIGIBILITY:
Inclusion Criteria:

* Diabetes
* Patients that are scheduled to undergo above knee amputation due to complications associated with diabetes

Exclusion Criteria:

* Minors

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects suffering from long standing diabetes and scheduled to undergo an above knee amputation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
ultrasonographic appearance | at examination before surgery
  There is outcome measure pe se. This is an observational study. We intend to study the ultrasonographic appearance of the sciatic nerve and compare this ultrasonographic appearance with the histologic appearance of the nerve. We know the nerve in diabetic neuropathy appears ultrasonographically different than a normal nerve. We just want to study the changed appearance of the nerve under ultrasound examination with the corresponding appearance of the nerve under the microscope.

CONTACTS AND LOCATIONS:
Overall Officials: Shashi B Bhatt, MD, Principal Investigator — University of Toledo
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States